CLINICAL TRIAL: NCT06863753
Title: The Effect of Kangaroo Mother Care on Breastfeeding Success in The Early Postpartum Period: Randomized Controlled Study
Brief Title: The Effect of Kangaroo Mother Care on Breastfeeding Success in The Early Postpartum Period
Acronym: Mother Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gülhan VAROL, Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MEU-HEM-GV-220
Record Dates: First submitted 2025-01-05; First posted 2025-03-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Kangaroo Mother Care
Keywords: Kangaroo mother care; Breastfeeding; Kangaroo care; Skin-to-skin contact
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Prospective, Clinical trial with randomized control
Who Masked: Outcomes Assessor
Masking Description: In a randomized controlled experimental study, the mothers participating in the study and the person who will perform the statistical analysis will be masked. The researcher will not be masked. It will not be explained to the mothers which group they are in and it will be stated that kangaroo mother care and breastfeeding training will be provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kangaroo mother care (Experimental): The practice will take place in the mother and baby's room. Mother and baby will be prepared for the practice. Kangaroo mother care will be provided once, when the service, mother and baby are available, and then the practice will be performed. For skin-to-skin contact, the newborn will be laid naked on the mother's bare chest in the prone position, the newborn's abdomen and chest will be in contact with the mother's skin. Subsequently, the newborn's head will be turned to the side so that the airway remains open. The newborn will stay in this position for at least 45 minutes.
  Interventions: Other: Kangoroo mother care
- Control (No Intervention): No intervention will be made to the control grup, only the data will be collected at the same time as the study group.

INTERVENTIONS:
Other: Kangoroo mother care — Kangaroo mother care will be practiced once, when the service, mother and baby are available, and then the training will be given. For skin-to-skin contact, the newborn will be laid naked on the mother's bare chest in the prone position, the newborn's abdomen and chest will be in contact with the mother's skin. Subsequently, the newborn's head will be turned to the side so that the airway remains open. The newborn will stay in this position for at least 45 minutes.
  Arms: Kangaroo mother care

SUMMARY:
The primary aim of this study was to determine the effect of kangaroo mother care on breastfeeding success in the early postpartum period. The secondary aim was to determine the effect of kangaroo mother care on the vital signs of the mother and the baby.

DETAILED DESCRIPTION:
From the selected sample, assignments to the intervention and control groups will be made by stratified block randomization method and randomizer.org website. Since it is predicted that mothers' previous breastfeeding experiences may affect breastfeeding success, mothers will be stratified in terms of the number of births (first vaginal birth/ two vaginal births). After stratification, block randomization will be performed and mothers will be assigned to the intervention and control groups with similar characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for mothers

  * Being over 18 years of age
  * Agree to participate in the survey (those who signed the Informed Consent Form)
  * Having had their first or second normal birth
  * Being literate
  * Having no communication problems
  * Being a singleton pregnancy
  * Having a gestational age of 37-42 weeks
  * Being open to communication and cooperation
  * Having an intact family unit
* Inclusion Criteria for Babies:

  * Birth weight 2500-4000 gr. between
  * Born by normal delivery
  * APGAR score of 7 and above at 1 and 5 minutes
  * No health problems or congenital anomalies
  * Born between 37 and 42 weeks of pregnancy

Exclusion Criteria:

* Exclusion Criteria for Mothers:

  * Being under 18 years of age
  * Do not agree to participate in the study
  * Not being able to read or write
  * Having more than two babies
  * Having breast problems that prevent breastfeeding
  * Being born by Caesarean section
  * Having a diagnosed mental or psychological disorder
* Exclusion Criteria for Babies:

  * Weighing less than 2500 grams
  * Weighing more than 4000 grams
  * Being born by Caesarean section
  * APGAR score of less than 7 at 1 and 5 minutes
  * Being born with a congenital anomaly
  * Born before 37 weeks

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who gave birth
Enrollment: 104 (Actual)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
LATCH Breastfeeding and Diagnostic Scale mean scores | Baseline and 60th minute
  This measurement tool consists of five items. The name of the diagnostic tool, LATCH, is formed from the first letters of these five criteria in English.
  * L, Latch on the breast;
  * A, Audible swallowing;
  * T, Type of the nipple;
  * C, Comfort breast/nipple of the mother;
  * H, Hold/Help position of the baby. Each item is evaluated between 0-2 points. The total score that can be obtained from the scale is 10, and a high score means high breastfeeding success.

SECONDARY OUTCOMES:
Vital signs of babies | Baseline and 60th minute
  Body temperature
Vital signs of mothers | Baseline and 60th minute
  Body temperature
Vital signs of babies | Baseline and 60th minute
  Respiratory rate
Vital signs of babies | Baseline and 60th minute
  Oxygen saturation
Vital signs of babies | Baseline and 60th minute
  Heart rate
Vital signs of mothers | Baseline and 60th minute
  Respiratory rate
Vital signs of mothers | Baseline and 60th minute
  Oxygen saturation
Vital signs of mothers | Baseline and 60th minute
  Heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin Hospital, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No